CLINICAL TRIAL: NCT02772497
Title: Three-month Outcome of Ziv-aflibercept for Diabetic Macular Edema
Brief Title: 3 Month Outcome of Ziv-aflibercept for DME
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Marashi Eye Clinic (Other)
Responsible Party: Principal Investigator, Ameen Marashi, MD, Marashi Eye Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol DME1
Record Dates: First submitted 2016-05-11; First posted 2016-05-13 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Anti VEGF; VEGF trap; Diabetes; Diabetic retinopathy; ZALTRAP; Ziv aflibercept
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ziv aflibercept (Experimental): Intravitreal ziv aflibercept 1.25 mg (0.05ml) every 4 weeks
  Interventions: Drug: Ziv aflibercept

INTERVENTIONS:
Drug: Ziv aflibercept — Intravitreal ziv aflibercept 1.25 mg (0,05ml) every 4 weeks
  Other Names: ZALTRAP

SUMMARY:
The purpose is to show the 3-month efficacy and safety in diabetic macular edema treated with intravitreal ziv-aflibercept.

DETAILED DESCRIPTION:
Multi-studies have shown that Intravitreal aflibercept (Eylea) is effective and safe in diabetic macular edema (DME) treatment and has gained FDA approval but it is expansive where ziv aflibercept (ZALTRAP) has the same molecule but with high osmilar buffer solution which is FDA approved for colon rectus cancer treatment and it is cost effective.

Studies have shown that intravitreal ziv aflibercept is safe and nontoxic despite the high osmolarity and even has short term effect in wet age related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with central diabetic macular edema
* Best corrected visual acuity is 20/25 or less
* Central macular thickness more than 250 microns
* Patients who are able to come for all follow-up

Exclusion Criteria:

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 3 years.
* Macular edema is present that is considered to be related to ocular surgery such as cataract extraction
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more
* History of major ocular surgery (including vitrectomy, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
* Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Proportion of visual acuity improvement using Snellen chart or equivalent | 3 months

SECONDARY OUTCOMES:
Amount of Central macular thickness reduction in microns after ziv-aflibercept treatment | 3 months
Amount of treatment cost in USD dollars | 3 months
Number of eyes with retinal toxicity after ziv aflibercept treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ameen Marashi, MD, Principal Investigator — Aleppo Syria

REFERENCES:
- [Result] Marashi A (2016) Three-Month Outcome of Ziv-Aflibercept for Diabetic Macular Edema. Adv Ophthalmol Vis Syst 4(3): 00114. DOI: 10.15406/aovs.2016.04.00114
- See also: Marashi A (2016) Three-Month Outcome of Ziv-Aflibercept for Diabetic Macular Edema. Adv Ophthalmol Vis Syst 4(3): 00114. DOI: 10.15406/aovs.2016.04.00114 — http://medcraveonline.com/AOVS/AOVS-04-00114.pdf